CLINICAL TRIAL: NCT04903275
Title: Caries Inhibition With CO2-Laser During Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MedicalUniversity_LaserCentre
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Caries; Initial
Keywords: carbon dioxide laser; fluoride; orthodontic treatment; caries inhibition
MeSH Terms: interventions — Fluoride Treatment

STUDY DESIGN:
Intervention Model Description: randomized, split-mouth controlled, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride and Laser (Experimental): In the split-mouth design, the left maxillary anterior teeth receive topical fluoride application and carbon dioxide (CO2) laser irradiation.
  Interventions: Procedure: Topical fluoride application and Laser irradiation
- Fluoride (Active Comparator): In the split-mouth design, this arm - the contralateral teeth (right maxillary incisors), will receive topical fluoride application.
  Interventions: Procedure: Topical fluoride application

INTERVENTIONS:
Procedure: Topical fluoride application and Laser irradiation — Topical fluoride varnish application (Clinpro™ White Varnish 5% Sodium Fluoride, 3M ESPE, USA) of the vestibular surfaces of the left maxillary anterior teeth followed by laser irradiation with CO2-laser (Ultra Dream Pulse, DS_40U, Daeshin Enterprise, Seoul, South Korea), emission wavelength 10,600 nm, time on-100 μs, time off-40 ms; average power-0.73 W; peak power-292.73 W; speed of movement-2 mm/s; energy density with movements-5 J/cm2; tip-to-tissue distance-20 mm; tip diameter 700 μm; irradiation time-30 s.
  Arms: Fluoride and Laser
Procedure: Topical fluoride application — Topical fluoride varnish application (Clinpro™ White Varnish 5% Sodium Fluoride, 3M ESPE, USA) of the vestibular surfaces of the left maxillary anterior teeth
  Arms: Fluoride

SUMMARY:
The aim of the study is to assess the viability and efficacy of carbon dioxide laser in combination with a fluoride varnish in the prevention, severity, and extent of white spot lesions during orthodontic treatment with fixed appliances.

DETAILED DESCRIPTION:
White spot lesions associated with orthodontic treatment are a common problem. The carbon dioxide laser is reported to be the most effective one in the prevention of dental caries. The study is designed as a randomized, split-mouth controlled, clinical trial. The participants will be children aged 12-18 years at high caries risk, requiring fixed orthodontic treatment. The vestibular surfaces of the maxillary anterior teeth of the eligible patients will be exposed to carbon dioxide laser irradiation in combination with fluoride therapy and fluoride therapy alone followed by bonding of orthodontic brackets. The patients will be recalled 6 and 12 months post-irradiation. Outcome measures will be visual examination with the International Caries Detection and Assessment System (ICDAS) criteria and SoproLife ® Daylight and Blue fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study are children ages 12 and older, in good general health
* Children, requiring fixed orthodontic treatment (brackets)
* Children at high caries risk according to 'Oral disease risk assessment tool' accepted and used in the Department of Paediatric Dentistry, Faculty of Dental medicine, Medical University - Plovdiv, Bulgaria
* Children with untreated non-carious vestibular surfaces of the six maxillary anterior teeth of the permanent dentition (central and lateral incisors, canines) with ICDAS code 0
* Verbal assent from the child willing to comply with all study procedures and protocol
* Obtained written informed consent by the patient's parent/guardian for participation in the study

Exclusion Criteria:

* Children with systemic diseases that may affect oral health or oral microflora (such as diabetes, etc.)
* Children with medication intake that could affect the salivary flow or oral microflora (such as antibiotics, etc.)
* Children with mental or cognitive problems
* Patients with maxillary anterior permanent teeth affected by disturbances in the development of dental structures (hypoplasia, hypomineralization, fluorosis)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes into International Caries Detection and Assessment System (ICDAS) codes | 1 year
  The International Caries and Detection System (ICDAS) is a visual scoring system developed for use in clinical assessment and clinical research of caries development and progression. It uses a numbered scoring system with a range from 0 to 6, to grade enamel demineralization and cavitation. Code of '0' represents unaffected/sound enamel, no caries change, '1' - first visual change, represents initial demineralization that is visible only after air drying, '2' represents a distinct visual change in the enamel that is visible when the surface is wet, '3' represents localized enamel loss or breakdown, no visible dentin or underlying shadow, and '4-6' represent larger carious lesions in dentin.

SECONDARY OUTCOMES:
Changes in SoproLife ® scores | 1 year
  The SOPROlife score is a visual assessment of the caries levels. The SoproLife ® daylight intraoral camera (SoproLife ® Daylight mode) is used to record an intraoral picture with Sopro-imaging software (Acteon, Sopro, La Ciotat, France). The SoproLife ® blue fluorescence mode scores range from 0 to 5. Code of '0' is given when the surface appears shiny green, the enamel appears sound, and there are no visible changes, code '1' - a tiny, thin red shimmer is observed, no red dots appeared, code '2' - darker red spots are visible, code '3' - dark red spots have extended, a slight beginning roughness of the red areas can be visible, and codes '4-6' represent larger carious lesions in dentin.

CONTACTS AND LOCATIONS:
Overall Officials: Ani B Belcheva, PhD, Study Director — Medical University Plovdiv, Bulgaria
Locations (2):
- Bulgaria (2):
  - Department of Paediatric Dentistry, Faculty of Dental Medicine, Medical University - Plovdiv, Bulgaria, Plovdiv
  - Medical University - Plovdiv, Bulgaria, Plovdiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belcheva AB, Shindova MP. Caries inhibition with CO2-laser during orthodontic treatment: a study protocol for a randomized split-mouth controlled clinical trial. Trials. 2022 Mar 12;23(1):208. doi: 10.1186/s13063-022-06117-y. PMID 35279220